CLINICAL TRIAL: NCT02361307
Title: The Outcomes of Seamless ADL Training Between Occupational Therapist and Nurse in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Poungkaew Thitisakulchai, Instructor, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Si 644/2014
Record Dates: First submitted 2015-01-28; First posted 2015-02-11 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional ADL training (Placebo Comparator): The control group receive the conventional ADL training programme
  Interventions: Procedure: Conventional ADL training
- seamless ADL training (Active Comparator): The experimental group receive the seamless ADL training programme which occupational therapist and nurse work with effective communication and cooperate in dressing and bathing training.
  Interventions: Procedure: Seamless ADL training

INTERVENTIONS:
Procedure: Seamless ADL training — The experimental group receive the seamless ADL training which occupational therapist and nurse work with effective communication and cooperate in dressing and bathing training
  Arms: seamless ADL training
Procedure: Conventional ADL training — The control group receive the conventional ADL training programme
  Arms: conventional ADL training

SUMMARY:
This study aimed to develop and implement an interdisciplinary team model with integration of all the relevant expertise and to establish powerful collaboration and communication among the team. To this extent, we designed a new approach toward self-care training called the "seamless self-care training" technique, which involves enhanced coordination and communication between OTs and nurses in the rehabilitation ward to promote interdisciplinary cooperation in self-care training.

DETAILED DESCRIPTION:
Rehabilitation is mandatory to promote functional recovery and minimize the distress of stroke survivors as much as possible. Even though rehabilitation outcomes are expected in all aspects, in one study the highest improvements were observed for bowel and bladder functions, transfer, and mobility, while the lowest improvements were seen in bathing (washing oneself), grooming (caring of body parts), dressing, and stair climbing.

Occupational therapists (OTs) are responsible for assessing and teaching skills to facilitate patients' activities and participation, including maximizing their performance of ADLs, and provide training programs and techniques that are tailor-made for each individual's impairment using targeted task-specific training, which has been acknowledged as the most effective method for enhancing functional outcomes. Nevertheless, the most important key factor for successful training outcomes is the collaboration of multiple healthcare professionals. All team members, especially nurses who spend lots of time with patients, should focus on encouraging and facilitating patients in transferring the newly relearned skills from professionals into their lives. Unfortunately, each expert usually approaches the patients from their own aspects, causing a lack of team perspective that could potentially preclude the patients from achieving their rehabilitation goals.

In current inpatient rehabilitation practice, there is still a gap in carrying out self-care training. Self-care training is usually carried out by OTs at the occupational therapy unit, whereas nursing staff assists washing and dressing the patients during admission at the rehabilitation ward. Due to time constraints, nurses usually concentrate on preparing the patients to be ready on time for other specific training. This hinders them from allowing patients the time and opportunity to practice by themselves, resulting in patients' having low confidence and a perception of low self-efficacy. Consequently, some patients may not develop sufficient skills to perform self-care independently after discharge. This situation was reported by Pryor and Long that an integrative function of nurses and other professionals was sub-optimal.

Therefore, in the present study, we aimed to develop and implement an interdisciplinary team model with integration of all the relevant expertise and to establish powerful collaboration and communication among the team. To this extent, we designed a new approach toward self-care training called the "seamless self-care training" technique, which involves enhanced coordination and communication between OTs and nurses in the rehabilitation ward to promote interdisciplinary cooperation in self-care training. We hope that this technique could make therapeutic intervention more successful and fill the gap in treatment processes, as well as to increase the self-efficacies of stroke survivors. The objective of this study was to explore the outcomes of providing this seamless self-care training to stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* First attack of stroke
* Good sitting balance
* TMSE 24 or more
* Need help in dresssing and bathing

Exclusion Criteria:

* Bilateral hemiparesis
* Dependent ADL before stroke attack
* Dementia
* Depression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Poungkaew Thitisakulchai, MD, Principal Investigator — Department of Rehabilitation Medicine
Locations (1):
- Poungkaew Thitisakulchai, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional ADL Training: The control group receive the conventional ADL training program
- Seamless ADL Training: The experimental group receive the seamless ADL training program which occupational therapist and nurse work with effective communication and cooperate in dressing and bathing training.
Period: Overall Study
Arm/Group | Conventional ADL Training | Seamless ADL Training
Started | 18 | 18
Completed | 18 | 17
Not Completed | 0 | 1
Not completed — Unstable medical condition. | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant in the experiment group discontinued the program due to a medical condition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional ADL Training | Seamless ADL Training | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (10.9) | 57.1 (10.3) | 58.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] | 18 | 17 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 18 | 17 | 35
Self-care score [Mean (Standard Deviation); unit: units on a scale] — Self-care score for dressing and washing oneself has minimum score of 0 for totally dependent performance and maximum score of 40 for the independent performance. These two activities consisted of 20 steps in total. Each step could be scored as 0, 1, or 2. A score of 2 meant the patients could perform the task independently, while 1 meant the patients could do the task with verbal cueing, and 0 meant the patients could not perform the task within 5 minutes or needed assistance to complete the task.
  units on a scale | 31.2 (7.6) | 29.6 (6.7) | 30.4 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Ability of Dressing and Bathing
Description: Normalized gain
  The raw score from the self-care checklist for dressing and washing oneself was used to calculate the normalized gain. Because stroke patients had varying scores for their initial dressing and washing oneself abilities, their possible window of improvement could be limited by the "floor to ceiling" effect. Therefore, it was considered that their improvements should be assessed by the normalized gain, which was introduced by Hake as a rough measure of the effectiveness of a training course and has since become the standard method for reporting scores. Hake defined normalized gain (g) as the ratio of the actual gain to the maximum possible gain as given in the equation:
  Normalized gain (g) = (post-training) - (pre-training) / (maximum score) - (pre-training) With a possible value between 0.0-1.0, the normalized gain can be divided into 3 levels: ''high-g'' for g ≥ 0.7, ''medium-g'' for 0.3 ≤ g ˂0.7, and ''low-g'' for g ˂ 0.3 The higher score means a better outcome.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Conventional ADL Training: The control group receive the conventional ADL training program
  Conventional ADL training: The control group receive the conventional ADL training program
- Seamless ADL Training: The experimental group receive the seamless ADL training programme which occupational therapists and nurse work with effective communication and cooperate in dressing and bathing training.
Arm/Group | Conventional ADL Training | Seamless ADL Training
Number analyzed (Participants) | 18 | 17
score on a scale | 0.71 (0.3) | 0.96 (0.1)
Statistical Analysis 1: Comparison: Conventional ADL Training vs Seamless ADL Training; Test type: Superiority; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Conventional ADL Training | Seamless ADL Training
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT02361307/Prot_SAP_000.pdf